CLINICAL TRIAL: NCT02415023
Title: A Phase Ib/2 Clinical Study to Evaluate the Safety, Pharmacokinetic Characteristics and Preliminary Efficacy of Fruquintinib Combined With Paclitaxel in Patients With Advanced Gastric Cancer
Brief Title: A Phase Ib/2 Clinical Study of Fruquintinib Combined With Paclitaxel in the Treatment of Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-013-00CH3
Record Dates: First submitted 2015-04-01; First posted 2015-04-14 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2018-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fruquintinib+paclitaxel (Experimental): fruquintinib combined with paclitaxel. Fruquintinib treatment: administration for 3 weeks followed by 1-week break, and administration every day for the first 21 days.Paclitaxel is administered once weekly in the first three weeks of each cycle.
  Interventions: Drug: fruquintinib+paclitaxel

INTERVENTIONS:
Drug: fruquintinib+paclitaxel — 28-day cycle of fruquintinib qd for 3 weeks followed by 1-week break combined with paclitaxel 80 mg/m2
  Other Names: HMPL-013+paclitaxel

SUMMARY:
An open-label, dose escalation and maximum tolerated dose (MTD) and/or recommended phase II dose (RPTD) study of fruquintinib combined with paclitaxel in patients with advanced gastric cancer who did not respond to first-line standard chemotherapy.

DETAILED DESCRIPTION:
In dose escalation period, 12-24 patients with advanced gastric cancer will be enrolled. Patients meeting enrollment eligibility will receive 28-day cycles of fruquintinib 2-5 mg qd combined with paclitaxel 80 mg/m2. Safety information and pharmacokinetic data will be collected till disease progression or intolerable toxicity to determine MTD and/or RPTD of fruquintinib combined with paclitaxel in patients with advanced gastric cancer. This period will include the following 4 dose groups from low to high:

A: Fruquintinib 2 mg qd for 3 weeks followed by 1-week break + paclitaxel 80 mg/m2 once a week during the first three weeks of each cycle B: Fruquintinib 3 mg qd for 3 weeks followed by 1-week break + paclitaxel 80 mg/m2 once a week during the first three weeks of each cycle C: Fruquintinib 4 mg qd for 3 weeks followed by 1-week break + paclitaxel 80 mg/m2 once a week during the first three weeks of each cycle D: Fruquintinib 5 mg qd for 3 weeks followed by 1-week break + paclitaxel 80mg/m2 once a week during the first three weeks of each cycle This study will use traditional 3+3 trial design (3 subjects will be enrolled in each dose group first. If 1 case of DLT is observed, additional 3 subjects will be enrolled in the same dose group to further evaluate toxicity) to observe DLT and evaluate MTD. If there are 2 or more cases of DLT in one dose group, the group lower than this dose group by one level is MTD dose group. At least 6 subjects are required in MTD dose group for confirmation. If MTD is not achieved at the end of dose escalation and there are 6 subjects in the highest dose group, RPTD can be determined based on obtained safety, tolerability, PK and efficacy information. Dose escalation and study in the next dose group can be initiated only after the first treatment cycle (DLT window observation period) is completed and subject safety and tolerability are confirmed in this dose group (0/3 or ≤1/6 subjects experience DLT).

Subjects in the original dose group will continue to receive the next cycle of treatment at the original dose till disease progression or treatment withdrawal due to any of the following reasons: 1) death, 2) intolerable toxicity, 3) pregnancy, 4) the investigator considers the study should be terminated for the subject's best interests, 5) the subject or legal representative requests withdrawal, 6) loss to follow-up, 7) the subject has poor compliance and cannot comply with the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study and sign the informed consent form voluntarily;
2. Patients with local advanced and/or metastatic gastric cancer confirmed by histology and/or cytology;
3. Fail in previous first-line standard chemotherapy
4. Aged 18-70years (inclusive);
5. Body weight ≥40 kg;
6. At least one measurable lesion (according to RECIST1.1);
7. Physical status score (ECOG score) 0-1;
8. Expected survival >12 weeks.

Exclusion Criteria:

1. Who are participating in another drug clinical trial in the past 4 weeks; or receive systemic anti-tumor chemotherapy, radiotherapy or biotherapy within 4 weeks prior to administration of the study drug;
2. Who previously received VEGF/VEGFR inhibitors;
3. Who have not recovered from toxicity caused by previous anti-cancer treatment (CTCAE>grade 1), or not completely recovered from previous surgery;
4. Active brain metastasis(with clinical symptom);
5. Other malignancies except squamous-cell or basal cell carcinoma, and cervical carcinoma in situ in the past 5 years;
6. Uncontrolled clinical active infection, e.g. acute pneumonia, hepatitis B or active hepatitis C;
7. Dysphagia, intractable vomiting or known drug malabsorption;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-11-09 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
incidence of DLT | every subject's DLT observation window is 4 weeks
progression free survival of RP2D | from first dose up to progressive disease or EOT due to any cause, assessed up to 1 year
  using RECIST v1.1 progressive disease (PD), using RECIST v 1.1
safety and tolerance | From first dose to within 30 days after the last dose
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 4.0.

SECONDARY OUTCOMES:
Objective response rate (ORR) | from first dose up to progressive disease or EOT due to any cause, assessed up to 1 year]
  using RECIST v 1.1
Disease control rate (DCR) | From first dose up to progressive disease or EOT due to any cause, assessed up to 1 year]
  using RECIST v 1.1
Pharmacokinetic profiles of Fruquintinib combined with Paclitaxel | From first dose up to day 15 in the first 28-day cycle
  PK sampling of Fruquintinibwill include a pre-dose and 1,2,4,8,24 hours time-point at Day 2 and day 15 of dosing in the first 28-day cycle; PK sampling of Paclitaxel will include a pre-dose and at 0.25,1,2,4,8, and 24 hours time-point on day 1 and day 15 of dosing in the first 28-day cycle

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Hutchison Medi Pharma Investigational Site, Beijing
  - Hutchison Medi Pharma Investigational Site, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] 1. The 16th Annual Meeting of Chinese Society of Clinical Oncology (CSCO) 2013 2. Elkerm YM, Elesaid A, AL-Batran, et al. Final results of a phase II trial of docetaxel-carboplatin- FU in locally advanced gastric carcinoma[abstract]. Presented at the 2008 gastrointestinal cancers symposium 2008.